CLINICAL TRIAL: NCT03365427
Title: Effect of Applications on Smart Phone on Post-operative Rehabilitation of Total Knee Arthroplasty: A Randomized Clinical Trail
Brief Title: Post-operative Rehabilitation of Total Knee Arthroplasty With Applications on Smart Phone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Lin Chutong, The clinical professor of arthritis clinic and research center, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PUPH20170917
Record Dates: First submitted 2017-12-02; First posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Osteoarthritis, Knee; Arthropathy of Knee
Keywords: rehabilitation; application on smart phones
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Application Group (Experimental): People in this arm will be introduced to an APP on smart phone, and receive lessons on how to use it on their own phones. The APP will be installed and prepare to use before surgery. People will be asked and monitored on-line to regularly use the APP.
  Interventions: Other: APP
- Convention Group (No Intervention): People in this arm receive exactly the same treatment and lessons on post-operative rehabilitation except the reach of the APP.

INTERVENTIONS:
Other: APP — An APP designed for patients experienced TKA, including on-line lessons on the action, frequency, intensity of rehabilitation exercises, and reporting system monitored by stuff from surgery team.
  Arms: Application Group

SUMMARY:
This study is designed to estimate the effect of an application on rehabilitation for osteoarthritis patients after total knee arthroplasty.

DETAILED DESCRIPTION:
Apart from surgical technique, the outcome of total knee arthroplasty (TKA) also largely depend on adequate rehabilitation and subsequent functional recovery after surgery.Rehabilitation affects or even determines various performance of post-operative knee, including knee range-of-motion (ROM), muscle strength, functional independence, all of which subsequently affect patients' quality of life. Conventional way of rehabilitation is exercise therapy, which rely on guidance of therapists and the self-efficacy of patients.

An application (APP) on smart phone was designed for people received TKA to play the role of guider and help improving patients' self-efficacy. This is a single-centre randomized clinical trial, with an anticipation of 200 patients with knee osteoarthritis enrolled, who will be randomly assigned into experiment group or control group. The patients in the experiment group will be introduced to this APP and requested to use it regularly, while the patients in the control group will receive pure conventional rehabilitation. Primary outcome includes Visual analogue scale (VAS) of pain, knee society score (KSS), ROM, ability of daily living (ADL) before operation and at 2 weeks and 6 weeks after surgery. All potential covariates of those two groups, such as age, sex, and pre-operative kellgren-lawrence scores would be matched by completely randomize.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as knee osteoarthritis with bearing X-ray
* Education level of middle school and above
* Prepared to take single-knee primary TKA

Exclusion Criteria:

* Severe varus/valgus (over 10 degree) of affected knee before surgery
* Stiffness of affected knee before surgery

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-01-07 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
The change of knee pain | before operation, 2 and 6 weeks after operation
  To use the Visual analogue scale (VAS) to estimate the pain of the affected knee. Its score ranges from 0 to 10, and higher score means more severe pain.

SECONDARY OUTCOMES:
The change of the range of motion of affected knee | before operation, 2 and 6 weeks after operation
  Use a goniometer to mesrange of motion of affected knee
The change of the symptoms of the affected knee | before operation, 2 and 6 weeks after operation
  To use the knee society score to estimate the symptoms of the affected knee.Its score ranges from 0 to 100, and higher score means more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jianhao Lin, MD, Principal Investigator — arthritis clinic and research center

IPD SHARING:
Plan to Share IPD: No